CLINICAL TRIAL: NCT05348291
Title: Ventilation Tubes for Recurrent Acute Otitis Media - Effects on Antibiotic Consumption and Otitis Media Episodes
Brief Title: Effect of Ventilation Tubes in Otitis-prone Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rorstudien2022
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Acute Otitis Media
Keywords: ventilation tubes; prevention; quality of life; antibiotic treatment; otitis media with effusion; audiometry; watchful waiting; tympanic membrane perforation
MeSH Terms: conditions — Otitis Media; Otitis Media with Effusion; Tympanic Membrane Perforation

STUDY DESIGN:
Intervention Model Description: Unblinded, randomised controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilation tubes (Active Comparator): Ventilation tube surgery
  Interventions: Device: ventilation tubes
- Active monitoring (No Intervention): Active monitoring of patients, with the possibility to cross over to other arm if deemed necessary.

INTERVENTIONS:
Device: ventilation tubes — Transtympanic pressure equalising devices.
  Other Names: grommets
  Arms: Ventilation tubes

SUMMARY:
The purpose of this study is to investigate the effects of ventilation tubes in children with recurrent ear infections. By drawing lots, young children with recurrent ear infections will be assigned to one of two groups (ventilation tubes or close follow-up), and the number of ear infections and antibiotic prescriptions in each group will be monitored. The study participants will be followed until they are 7 years old.

DETAILED DESCRIPTION:
Children who fulfil the criteria of recurrent acute otitis media (AOM) before they are one year of age will be randomised to ventilation tube surgery or active monitoring (50% vs 50%). Due to the nature of the intervention, blinding will not be possible. Children randomised to are randomised to active monitoring and continue to have frequent recurrences will be given the opportunity to cross between groups.

Children will be followed by the study doctors every third month until the age of two years, and after this yearly. In addition to planned visits, the families will be advised to contact the study doctors whenever they suspect that their child has a new episode of AOM. Otomicroscopy and nasopharyngeal cultures will be performed at every visit; cultures from the external ear canal will be taken when applicable. It will also be noted whether there is any perforation of the tympanic membrane, whether ventilation tubes are still in place, whether there is an ongoing episode of AOM or of otitis media with effusion (OME). At each planned visit, a parental quality of life questionnaire for children with ear disease will be completed. It will be noted how many AOM episodes the child has had since the last planned visit, how many times the patient has been prescribed oral antibiotics (also for reasons other than AOM), and if the family has seen a doctor elsewhere. At each emergency visit, it will be noted if the child has AOM or not, whether the child has fever, any signs of complications to AOM, a spontaneous perforation and whether the child´s general well-being is affected.

At the ages of 4 and 7 years and, if a hearing impairment is suspected on any other occasion, hearing tests will be performed.

ELIGIBILITY:
Inclusion Criteria: At inclusion, children should be under 1 year of age and fulfil the internationally accepted definition of recurrent AOM, ie have had 3 episodes of AOM during the last 6 months, or 4 during the last 12 months.

-

Exclusion Criteria: chromosomal aberrations, cleft palate or severe immune deficiency

-

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Antibiotic prescriptions | First two years in study
  Number of oral antibiotic prescriptions
Otitis media episodes | First two years in study
  Number of otitis media episodes

SECONDARY OUTCOMES:
Microbiology | First two years in study
  Nasopharyngeal and middle ear growth during acute otitis media episodes
Tympanic membrane perforations | Until age 7
  Presence of chronic tympanic membrane perforations
Audiometry | At age 4 and 7 years
  Audiometry, including high frequency audiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery, Lund, Sweden